CLINICAL TRIAL: NCT00711399
Title: Use of Objective Cough Counting and Breath Sounds Documenting Device, to Assess the Severity and Duration of Cough and Wheeze in Children and Adults Suffer From Acute or Chronic Respiratory Disease.
Brief Title: Assessment of Cough and Wheeze With Breath Sound Documenting Device
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Haim Bibi MD, Carmel Medical Center
Other Study IDs: CMC 07-0063
Record Dates: First submitted 2008-06-18; First posted 2008-07-08 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Respiratory Sounds
Keywords: Respiratory sounds; Wheeze; Cough
MeSH Terms: conditions — Respiratory Sounds; Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- group A: Study group
  Interventions: Device: PulmoTrack® 2010 with WIM-PC™ and WIM-CC™ Technologies

INTERVENTIONS:
Device: PulmoTrack® 2010 with WIM-PC™ and WIM-CC™ Technologies — wheeze and cough detection in hospitalized patients.

SUMMARY:
The study goal is to create a database of respiratory sounds recordings, to evaluate and validate the WIM technology and to evaluate the efficacy of a specific treatment by comparing the severity of the respiratory symptoms before and after the administration of the treatment.

DETAILED DESCRIPTION:
Clinical background Respiratory wheezes are a characteristic symptom of asthma and other obstructive diseases. The wheezes can be heard on the chest surface and on the trachea using a stethoscope or by listening near the person's mouth. The wheezes are a part of the Continuous Adventitious Breath Sounds (CABS) family, in addition to the wheezes, the rhonchi and the whistles are also a part of this family. Each breath sound has its own unique characteristics but all of them indicate a presence of an airway obstruction. Reducing the obstruction by bronco dilators, for example, lowers the amount of wheezes; meaning lowers the time period during the breathing when wheeze is present.

Cough is part of the defense mechanism to protect the lung from foreign particles and remove secretions from the airways. However, at times it becomes a bothersome, annoying symptom that interferes with the quality of life, sleep pattern and exercise tolerance of the patient.

Children with respiratory infection, asthmatic children and CF patients suffer from a multitude of pathologies of airways and are often inflicted with chronic cough.

Recently a breakthrough in continuous monitoring of respiratory symptoms was introduced. The Wheezing Infant Monitor (WIM) is a technology that utilizes a flat coin shape microphone that is attached to the chest and over the trachea and allows a continuous recording of the breath sounds absorbed by the microphone. This innovative technology provides an objective assessment of the duration, intensity and timing of the respiratory symptoms after a computerized processing of the data.

Study background The study title is 'Use of objective cough counting and breath sounds documenting device, to assess the severity and duration of cough and wheeze in children and adults suffer from acute or chronic respiratory disease'. The study goal is to create a database of respiratory sounds recordings, to evaluate and validate the WIM technology and to evaluate the efficacy of a specific treatment by comparing the severity of the respiratory symptoms before and after the administration of the treatment.

The study is an open study. Each patient will be evaluated twice during each day of hospitalization. Each recording session will last about one hour and include 10 minutes of pre treatment recording, administration of the treatment and continuation of the recording. The patient will be treated according to his/her condition and the recording will not delay the administration of the treatment in urgent cases.

The study population will consist of children with respiratory infection, asthmatic children and CF patients who suffer from respiratory symptoms such as cough and/or shortness of breath. The study population will include approximately 200 patients.

Patients with cough, wheeze or shortness of breath and patients (or their parents/guardians) who gave their consent to participate in the study will be included. Subjects who are in respiratory distress, have skin lesions precluding attachment of sensors, subject with chest tubes and pregnant women will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient and/or parents/guardian signed informed consent
* Patients with cough or shortness of breath

Exclusion Criteria:

* Chest tubes
* Skin lesions precluding attachment of sensors
* Respiratory distress
* Pregnant women

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of children with respiratory infection, asthmatic children and CF patients who suffer from respiratory symptoms such as cough and and/or shortness of breath.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Respiratory sounds recordings | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Goryachev, BSc, Study Chair — KarmelSonix Ltd.
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- See also: Breath sound recorder WIM-PC™ — http://www.karmelsonix.com